CLINICAL TRIAL: NCT04392258
Title: Observational and Diagnostical Study on Transient Allostatic Responses of Thyroid Function After Cardiopulmonary Resuscitation
Acronym: Thyro-CPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, PD Dr. Johannes W. Dietrich, MD, Consultant endocrinologist, Ruhr University of Bochum
Other Study IDs: 19-6678-BR; U1111-1251-7468 (Other: WHO Universal Trial Number (UTN)); DRKS00021695 (Registry Identifier: Deutsches Register Klinischer Studien / German Clinical Trials Register (DRKS))
Record Dates: First submitted 2020-05-07; First posted 2020-05-18 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Heart Arrest; Ventricular Fibrillation; Ventricular Flutter; Ventricular Tachycardia
Keywords: thyroid; homeostasis; allostasis; resuscitation; allostatic load; critical illness; TACITUS; NTIS; Circulatory arrest
MeSH Terms: conditions — Heart Arrest; Ventricular Fibrillation; Ventricular Flutter; Tachycardia, Ventricular; Thyroid Diseases; Critical Illness | interventions — Thyroid Function Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum aliquots are stored for postponed determination of non-classical thyroid hormones including but not limited to thyronamines, 3,5-diiodothyronine (3,5-T2) and reverse T3 (rT3).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Status post resuscitation: Patients or dataset that underwent resuscitation
  Interventions: Diagnostic Test: TSH determination; Diagnostic Test: FT4 determination; Diagnostic Test: FT3 determination; Diagnostic Test: SPINA-GT; Diagnostic Test: SPINA-GD

INTERVENTIONS:
Diagnostic Test: TSH determination — Determination of serum concentration of thyrotropin (TSH)
  Other Names: serum thyrotropin determination
Diagnostic Test: FT4 determination — Determination of serum free thyroxine (FT4) concentration
  Other Names: serum free T4 determination
Diagnostic Test: FT3 determination — Determination of serum free triiodothyronine (FT3) concentration
  Other Names: serum free T3 determination
Diagnostic Test: SPINA-GT — Calculation of thyroid's secretory capacity (SPINA-GT)
  Other Names: GT; Thyroid's secretory capacity; LOINC 82368-2; thyroid's incretory capacity
Diagnostic Test: SPINA-GD — Calculation of total deiodinase activity (SPINA-GD)
  Other Names: GD; Sum activity of peripheral deiodinases; LOINC 82367-4; deiodination capacity

SUMMARY:
Time-limited adaptive responses of thyroid function are common in the critically ill. About 70% of all patients treated on intensive care units develop a so-called non-thyroidal illness syndrome (NTIS) or TACITUS (thyroid allostasis in critical illness, tumours, uraemia and starvation), which is marked by low serum concentrations of the thyroid hormone T3 and other adaptive reactions of thyroid homeostasis. Occasionally, temporarily elevated concentrations of thyrotropin (TSH) and peripheral thyroid hormones are to be observed, especially after cardiopulmonary resuscitation (CPR). However, the available evidence is limited, although abnormal concentrations of thyroid hormones after CPR have occasionally been reported.

Aim of the planned study is to investigate the thyrotropic (i.e. thyroid-controlling) partial function of the anterior pituitary lobe immediately after CPR. It is intended to evaluate statistical measures of TSH concentration and peripheral thyroid hormones in de-identified datasets (protocol A). Additionally, a prospective sub-study (protocol B) aims at a more precise description of pituitary and thyroid responses by means of serial investigations in routine serum samples, both immediately after CPR and during the course of ongoing treatment. This includes the evaluation of additional possible predictors, too.

Primary endpoint of the study is changed TSH concentration immediately after CPR compared to the TSH value 24 hours later. Secondary endpoint is the relation between thyroid-controlling pituitary function and mortality.

A high proportion of patients undergoing CPR will eventually receive iodinated radiocontrast media (e.g. for computed tomography or coronary angiography). This is one of the reasons why early identifying subjects at high risk for possible iodine-induced thyrotoxicosis is important. Increased oxygen consumption of the heart in hyperthyroidism is one of the reasons for high mortality in thyrotoxicosis. Therefore, accurate diagnosis of alterations in the hypothalamus-pituitary-thyroid (HPT) axis is of paramount importance.

DETAILED DESCRIPTION:
Transient allostatic responses of thyroid function are common in the critically ill. About 70% of all patients treated on intensive care units develop a so-called non-thyroidal illness syndrome (NTIS) or TACITUS (thyroid allostasis in critical illness, tumours, uraemia and starvation), which is marked by low serum concentrations of the thyroid hormone T3 and other adaptive reactions of thyroid homeostasis. Occasionally, temporarily elevated concentrations of thyrotropin (TSH) and peripheral thyroid hormones are to be observed, especially after cardio-pulmonary resuscitation (CPR). However, the available evidence is limited, although abnormal concentrations of thyroid hormones after CPR have been reported.

Aim of the planned study is to investigate the thyrotropic partial function of the anterior pituitary lobe immediately after CPR. It is intended to evaluate statistical moments of TSH concentration and peripheral thyroid hormones in de-identified datasets (protocol A). Additionally, a prospective substudy (protocol B) aims at a more precise description of pituitary and thyroid responses by means of serial investigations in routine serum samples, both immediately after CPR and during the course of ongoing in-patient treatment. This also includes the evaluation of additional possible predictors.

Primary endpoint of the study are changed TSH concentrations immediately after CPR compared to the value 24 hours later. Secondary endpoint is the relation between thyrotropic pituitary function and mortality.

A high proportion of patients undergoing CPR will eventually receive iodinated radiocontrast media (e.g. for computed tomography or coronary angiography). This is one of the reasons why early identifying subjects at high risk for possible iodine-induced thyrotoxicosis is important. Increases oxygen consumption of myocardial tissue in hyperthyroidism is one of the reasons for high mortality in thyrotoxicosis. Therefore, accurate diagnosis of alterations in the hypothalamus-pituitary-thyroid (HPT) axis is of paramount importance.

ELIGIBILITY:
Inclusion Criteria:

* Admission after cardiopulmonary resuscitation
* Minimum age of 18 years
* Results of TSH and peripheral thyroid hormone concentrations already available or possibility to reorder these investigations in a post-hoc manner if consent has been obtained (i. e. time interval after venipuncture within the storage period of the central laboratory)
* Inclusion after own consent of the patient after reawakening, via custodian or independent consultant.

Exclusion Criteria:

* Missing data on thyroid homeostasis in the first blood specimen (obtained before 3 hours after admission)
* Traumatic brain injury
* Persistent hints for thyroid dysfunction, not explained by non-thyroidal illness syndrome (NTIS) / euthyroid sick syndrome (ESS) / thyroid allostasis in critical illness, tumors, uremia and starvation (TACITUS) in consecutive investigations over several days after resuscitation
* Functionally relevant thyroid or pituitary disorder, as documented in international classification of diseases (ICD) codes.
* Exposure to radiocontrast agents less than 3 months ago
* Therapy with amiodarone (currently or during the previous 3 years)
* Pregnancy
* Known thyroid disease
* Consent not obtained within the routine storage period of the central laboratory
* Post-hoc-exclusion if evidence for true dysfunction the the pituitary or the thyroid became available during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: De-identified datasets (protocol A) or patients (protocol B) admitted to an intensive care unit after cardiopulmonary resuscitation (CPR)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
TSH response | three hours
  Changes in TSH concentration after CPR compared to the value after 24 hours

SECONDARY OUTCOMES:
Prognosis | Through study completion, an average of 1 year
  Mortality dependent on pituitary thyrotropic partial function

CONTACTS AND LOCATIONS:
Overall Officials: Johannes W Dietrich, M.D., Principal Investigator — Bergmannsheil University Hospitals
Locations (1):
- Medizinische Klinik I, Universitätsklinikum Bergmannsheil, Ruhr-Universität Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Sharing may be considered upon reasonable request.

REFERENCES:
- [Background] Dietrich JW, Stachon A, Antic B, Klein HH, Hering S. The AQUA-FONTIS study: protocol of a multidisciplinary, cross-sectional and prospective longitudinal study for developing standardized diagnostics and classification of non-thyroidal illness syndrome. BMC Endocr Disord. 2008 Oct 13;8:13. doi: 10.1186/1472-6823-8-13. PMID 18851740
- [Background] Dietrich JW, Landgrafe G, Fotiadou EH. TSH and Thyrotropic Agonists: Key Actors in Thyroid Homeostasis. J Thyroid Res. 2012;2012:351864. doi: 10.1155/2012/351864. Epub 2012 Dec 30. PMID 23365787
- [Background] Dietrich JW, Muller P, Schiedat F, Schlomicher M, Strauch J, Chatzitomaris A, Klein HH, Mugge A, Kohrle J, Rijntjes E, Lehmphul I. Nonthyroidal Illness Syndrome in Cardiac Illness Involves Elevated Concentrations of 3,5-Diiodothyronine and Correlates with Atrial Remodeling. Eur Thyroid J. 2015 Jun;4(2):129-37. doi: 10.1159/000381543. Epub 2015 May 23. PMID 26279999
- [Background] Dietrich JW, Landgrafe-Mende G, Wiora E, Chatzitomaris A, Klein HH, Midgley JE, Hoermann R. Calculated Parameters of Thyroid Homeostasis: Emerging Tools for Differential Diagnosis and Clinical Research. Front Endocrinol (Lausanne). 2016 Jun 9;7:57. doi: 10.3389/fendo.2016.00057. eCollection 2016. PMID 27375554
- [Background] Chatzitomaris A, Hoermann R, Midgley JE, Hering S, Urban A, Dietrich B, Abood A, Klein HH, Dietrich JW. Thyroid Allostasis-Adaptive Responses of Thyrotropic Feedback Control to Conditions of Strain, Stress, and Developmental Programming. Front Endocrinol (Lausanne). 2017 Jul 20;8:163. doi: 10.3389/fendo.2017.00163. eCollection 2017. PMID 28775711
- [Background] Muller P, Dietrich JW, Lin T, Bejinariu A, Binnebossel S, Bergen F, Schmidt J, Muller SK, Chatzitomaris A, Kurt M, Gerguri S, Clasen L, Klein HH, Kelm M, Makimoto H. Usefulness of Serum Free Thyroxine Concentration to Predict Ventricular Arrhythmia Risk in Euthyroid Patients With Structural Heart Disease. Am J Cardiol. 2020 Apr 15;125(8):1162-1169. doi: 10.1016/j.amjcard.2020.01.019. Epub 2020 Jan 29. PMID 32087999
- [Background] Aweimer A, El-Battrawy I, Akin I, Borggrefe M, Mugge A, Patsalis PC, Urban A, Kummer M, Vasileva S, Stachon A, Hering S, Dietrich JW. Abnormal thyroid function is common in takotsubo syndrome and depends on two distinct mechanisms: results of a multicentre observational study. J Intern Med. 2021 May;289(5):675-687. doi: 10.1111/joim.13189. Epub 2020 Nov 12. PMID 33179374